CLINICAL TRIAL: NCT06070181
Title: "Effectiveness of Emdogain® As an Adjunctive Therapy for Non-Surgical Periodontal Treatment- a Randomized, Controlled, Split-Mouth Design Multicenter Clinical Trial"
Brief Title: Effectiveness of Adjunctive Therapy of Emdogain®FL in Non-surgical Periodontal Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ostergotland County Council, Sweden (Other)
Collaborators: Region Jönköping County (Other Government)
Responsible Party: Principal Investigator, Shariel Sayardoust, Associate professor and Senior Consultant in Periodontology, Ostergotland County Council, Sweden
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EMDFL2023
Record Dates: First submitted 2023-09-30; First posted 2023-10-06 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Periodontitis
Keywords: non-surgical treatment; Periodontal treatment; Periodontitis stage 3 and 4; Enamel matrix derivate; Emdogain flapless
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- Control- no adjunctive treatment (Other): One arm is the control: two quadrants per each patient treated with non-surgical periodontal treatment alone. NO adjunctive treatment with emdogain. The two quadrants are randomized.
  Interventions: Procedure: Non-surgical periodontal treatment
- Test-adjunctive treatment with Emdogain (Experimental): The experimental arm is the two quadrants per patient assigned to be treated vid adjunctive Emdogain.
  Interventions: Device: Enamel matrix derivate; Procedure: Non-surgical periodontal treatment

INTERVENTIONS:
Device: Enamel matrix derivate — 'Applying Enamel matrix derivate in the periodontal pockets after completing the non-surgical periodontal treatment
  Other Names: Emdogain
  Arms: Test-adjunctive treatment with Emdogain
Procedure: Non-surgical periodontal treatment — No additional/adjunctive treatment with Emdogain
  Other Names: Control- no adjunctive treatment

SUMMARY:
The goal of this clinical trial is to assess the safety and effectiveness of adjunctive Emdogain® therapy in non-surgical periodontal treatment for patients with stage 3 and 4 periodontitis.

The main questions it aims to answer are:

* Will adjunctive treatment with Emdogain® result in a greater reduction in Bleeding on Probing and probing pocket depth compared to non-surgical periodontal treatment alone? • Will adjunctive treatment with Emdogain® lead to a greater mean Radiographic attachment level (rAL) gain per quadrant compared to non-surgical periodontal treatment alone?
* Will adjunctive treatment with Emdogain® result in a lower proportion of treated teeth requiring surgery (PPD ≥6mm) at 12 months after treatment?

Participants in the study will undergo the following tasks:

* Screening and randomization
* Receival of non-surgical periodontal treatment in all quadrants and in two quadrants adjunctive Emdogain®
* 6-month follow-up assessment
* 12-month follow-up assessment

Clinical and radiological assesment will be performed in two quadrants treated with adjunctive Emdogain® therapy and two quadrants treated with non-surgical periodontal treatment alone. This comparison will help determine the effects of adjunctive therapy with Emdogain®.

The study aims to provide insights into the safety and efficacy of adjunctive Emdogain® therapy in non-surgical periodontal treatment, specifically in patients with stage 3 and 4 periodontitis.

DETAILED DESCRIPTION:
Phase 1: Screening After written informed consent has been obtained, the patient is entered in the screening and enrolment log and in the patient identification log and receives a patient identification number. An evaluation is then carried out by a periodontist with a dental hygienist to determine whether the patient meets the study inclusion criteria and none of the exclusion criteria and study specific information will be collected. For excluded patients, the reason(s) for exclusion shall be documented.

Phase 2: Treatment After providing informed consent, screening completion and after examination by a periodontist, study treatment will be performed only once the Plaque Index (PI) of each screened patient will be <20%. This means that randomization and the scaling phase (study treatment) will be only initiated when each individual patient was compliant with the oral hygiene instructions and the PI (as measured with Staining rondells red Directa, 4 surface plaque index, 1 rinsing 10 sec with 50 ml of water) was recorded to be <20%.

Randomization to test or control-quadrants will be performed using statistical software after full mouth scaling and root planing has taken place. Out of the four quadrants / patient, two quadrants will be randomised to be treated according to standard care with adjunctive Emdogain® FL. The remaining two quadrants will be treated as controls (standard care; no adjunctive Emdogain® FL).

Following randomization, root planing and scaling will be performed by a calibrated dental hygienist in all quadrants under local anaesthesia (with xylocaine adrenaline 2%). First, an ultrasonic scaler (EMS) will be used and then manual scaling with LM-curettes will be performed. The hygienist will scale each root surface until the root surface is judged to be free of tartar. As part of standard care, this decision is made by the calibrated dental hygienist based on tactile experience.

Pockets of 5mm to 9mm (PPD) will be treated in the study (both Test and Control treatment). Test treatment: Emdogain® FL will be added to standard treatment i. e. Test quadrants. PrefGel® will be applied on the root surface for 2 minutes, then rinsed away with sterile saline solution for 30 seconds. The surface will be lightly dried using gauze and airblow and then Emdogain® will be applied. The Emdogain® FL application will be performed by the dental hygienist under the supervision of a periodontist. Control treatment: pockets of 5mm to 9mm (PPD) will receive standard treatment (no addition of Emdogain® FL) i. e. Control quadrants.

Additional teeth with PPD outside the range of 5mm to 9mm (PPD) may be present both in Test and/or Control quadrants. Such teeth will be treated using standard care (no Emdogain®) but they will not be included in study evaluations.

The patient will then be asked to rinse daily with an antiseptic mouth rinse twice a day (FLUX-CHX chlorhexidine 0.12% solution) until 14 days following the treatment. Antibiotics (e.g. penicillin V) may also be used in the presence of suppuration. The patient will be instructed not to brush in the treated area for 7 days following the treatment. Then only gentle brushing on buccal and lingual tooth surfaces using the roll stroke method will be recommended. The patients will be instructed not to perform any sulcular or interdental brushing before 2 weeks following the treatment.

Followed by individually planed healing controls and oral hygiene controls. (the number of visits/follow-ups will be recorded and presented.

Phase 3: 6 months follow up Examination will be carried out by a periodontist (blinded) at the six months follow up visit. Examination consists of periodontal assessments i. e. PI, BoP and PPD.

Phase 4: 12 months follow up Examination will be carried out by a periodontist (blinded) at the 12 months follow up visit. Examination consists of periodontal assessments (PI, BoP, PPD) and X-rays.

ELIGIBILITY:
Inclusion Criteria:

Study Population The study population will consist of patients affected by Stage 3 or 4 periodontitis. See below for a full list of inclusion and exclusion criteria.

Inclusion Criteria

Patients must meet all of the following criteria for inclusion in the study:

* Over 18 years old
* Stage 3 or 4 periodontitis
* Residual pockets with probing depths from 5mm to 9mm with no furcation involvement and adequate plaque control

Exclusion Criteria:

Patients who meet any of the following exclusion criteria are not allowed to be included in the study:

* Antibiotic treatment in last 3 months
* Subgingival scaling and root planning performed in last 12 months
* Patients for which the use of Emdogain® is contraindicated i. e. patients with uncontrolled diabetes or other uncontrolled systemic diseases, disorders or treatments that compromise wound healing, chronic high dose steroid therapy, bone metabolic diseases, radiation or other immuno-suppressive therapy and infections or vascular impairment at the surgical site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Pocket Probing Depth (PPD) | baseline (before treatment), at 6 month and 12 moth after treatment
  The PPD will be measured around each tooth by recording the distance in millimeters (mm) from the gingival margin to the bottom of the pocket at 4 locations (mesial, buccal, distal, and palatal). The mean across all teeth within each quadrant will be determined.

SECONDARY OUTCOMES:
Changes in Proportion of sites with Bleeding on Probing (BoP) | baseline (before treatment), at 6 month and 12 moth after treatment
  BoP will be recorded. The presence or absence of BoP will be documented as a "yes" or "no" on 4 sites (mesial, buccal, distal, and palatal) around the tooth. The endpoint will be defined as the proportion of sites with BoP .
Mean rAttanchment Level (rAL) changes per quadrant | baseline (before treatment), and 12 moth after treatment
  Mesial and distal rAL will be recorded as the result of quantitative assessment of the standardized peri-apical / bite wing x-ray (by a qualified and validated blinded radiologist).
  For rAL assessment standardized peri-apical radiographs are taken at the time points listed in Table 2 i. e. at Visits 2 (after treatment) and 4 (12 months). Parallel technique will be used, with vertical bite wings for molars and premolars and peri-apical X-rays will be performed for incisors and canines.
Proportion of teeth which are indicated for surgery (PPD ≥ 6mm) at 12 months after treatment | 12 month after treatment
  Proportion of teeth with PPD ≥ 6mm at the 12 month follow up will be determined.

OTHER OUTCOMES:
Changes in the PI (Plaque Index) at 6 months and 12 months after treatment | baseline (before treatment), at 6 month and 12 moth after treatment
  PI will be recorded . The presence of plaque will be documented as "yes" or "no" on four sites (mesial, buccal, distal and palatal) around the tooth. The endpoint will be calculated as proportion of surfaces with plaque.

CONTACTS AND LOCATIONS:
Overall Officials: Shariel Sayardoust, PhD, DDS, Principal Investigator — Ostergotland County Council, Sweden
Locations (1):
- Centre for Oral Rhabilitation, Linköping, Region Östergötland, Sweden

IPD SHARING:
Plan to Share IPD: No